

# STATISTICAL ANALYSIS PLAN

#### LA38-EXT

Long-term Safety and Efficacy Study of Ferriprox® for the Treatment of Transfusional Iron Overload in Patients with Sickle Cell Disease or Other Anemias

Final Version 1.0

14 JUNE 2019

Prepared by

David Lee PhD

Scientific Leader, Biostatistics

ApoPharma Inc.

### **APPROVALS**

Caroline Fradette, PhD

Carol fr

Director of Clinical Research, ApoPharma Inc.

14 Lun 2019

Date (DD MMM YYYY)

Anna Rozova, MD

Director of Medical Safety, ApoPharma Inc.

14 Jun 2019

Date (DD MMM YYYY)

Yu Chung Tsang, PhD

Chief Scientific Officer, Biopharmaceutics &

Biostatistics, Apotex Inc.

14 Jan 2011 Date (DD MMM YYYY)

# TABLE OF CONTENTS

| <b>A</b> l | PPROVAL | S | 2 |
|------------|---------|------------------------------------|----|
| L | | BBREVIATIONS AND DEFINITIONS OF | |
| 1 | INTR | RODUCTION | 7 |
| 2 | STUD | DY OBJECTIVES | 7 |
| | 2.1 Pri | mary Objective | 7 |
| | 2.2 Sec | condary Objective | 7 |
| 3 | STUE | DY DESIGN | 7 |
| 4 | STUE | DY PROCEDURES | 7 |
| | 4.1 Me | ethod of Assignment to Treatment | 10 |
| | 4.2 Bli | nding Procedures | 10 |
| | 4.3 All | location of Patient Numbers | 10 |
| | 4.4 Tre | eatment Compliance | 10 |
| 5 | MEA | SUREMENTS AND EVALUATIONS | 10 |
| | 5.1 Eff | ficacy Measurements | 10 |
| | 5.1.1 | Liver Iron Concentration | 10 |
| | 5.1.2 | Cardiac MRI T2* | 10 |
| | 5.1.3 | Serum Ferritin | 10 |
| | 5.2 Saf | fety Measurements | 11 |
| | 5.2.1 | Adverse Events | 11 |
| | 5.2.2 | Serious Adverse Events | 11 |
| | 5.2.3 | Adverse Events of Special Interest | 11 |
| | 5.2.3 | 3.1 Neutropenia | 11 |
| | 5.2.3 | 3.2 Infections | 12 |
| | 5.2.4 | Laboratory Measurements | 12 |
| | 5.2.5 | Other Safety Measurements | 13 |
| | 5.2.5 | 5.1 Physical Examination | 13 |
| | 5.2.5 | 5.2 Vital Signs | 13 |
| | 5.2.5 | 5.3 Electrocardiogram | 13 |
| | 5.2.5 | 5.4 Concomitant Medications | 13 |
| 6 | STAT | TISTICAL ANALYSIS | 13 |
| | 6.1 End | dpoints | 13 |

| 611 | Primary Endpoints | 13 |
|---------|---------------------------------------|----|
| 6.1.2 | Secondary Endpoints | 14 |
| 6.2 Stu | dy Populations | 14 |
| 6.2.1 | Intent-to-Treat Population | 15 |
| 6.2.2 | Per Protocol Population | |
| 6.2.3 | Safety Population | 15 |
| 6.3 Da | ta Analysis | 15 |
| 6.3.1 | Patient Disposition and Drug Exposure | |
| 6.3.2 | Patient Characteristics | 15 |
| 6.3.3 | Analysis of Efficacy | 15 |
| 6.3.4 | Analysis of Safety | |
| 14 SUM | MARY TABLES AND FIGURES | |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| AE | Adverse event |
| AF | Assent form |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| CS | Clinically significant |
| CI | Confidence interval |
| CRA | Clinical research associate |
| CRF | Case report form |
| CRO | Contract research organization |
| DFO | Deferoxamine |
| DFP | Deferiprone |
| dw | Dry weight |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GGT | Gamma-glutamyl transferase |
| Hb | Hemoglobin |
| HIV | Human immunodeficiency virus |
| HR | Heart rate |
| ICF | Informed consent form |
| ICH | International Conference on Harmonisation |
| ID | Identification |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| ITT | Intent-to-treat |
| LIC | Liver iron concentration |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligram |
| mg/g | milligram per gram |
| NCS | Not clinically significant |

| Abbreviation | Definition |
|--------------|-------------------------------------|
| OCRDC | Oracle Clinical Remote Data Capture |
| PDR | Patient Data Report |
| PP | Per protocol |
| RBC | Red blood cell |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SCD | Sickle cell disease |
| t.i.d. | three times daily |
| ULN | Upper limit of normal |
| WHO | World Health Organization |

### 1 INTRODUCTION

This document outlines the statistical analysis plan (SAP) for LA38-EXT, titled "Long-term Safety and Efficacy Study of Ferriprox® for the Treatment of Transfusional Iron Overload in Patients with Sickle Cell Disease or Other Anemias".

Once patients in LA38-0411 have completed the study, they have been invited to enroll in LA38-EXT, a 2-year extension study in which all patients have received deferiprone. The long-term data obtained from this study will provide additional information on the safety and efficacy of deferiprone in patients with sickle cell disease or other anemias.

#### 2 STUDY OBJECTIVES

### 2.1 Primary Objective

To evaluate the long-term safety and tolerability of deferiprone in iron-overloaded patients with sickle cell disease or other anemias.

# 2.2 Secondary Objective

To evaluate the efficacy of deferiprone in the treatment of iron overload in patients with sickle cell disease or other anemias who have received deferiprone for up to 3 years.

#### 3 STUDY DESIGN

LA38-EXT is a 2-year prospective, multi-center, single-arm, open-label extension of LA38-0411. All patients who have completed LA38-0411 have been offered the opportunity to continue in this extension study, with the final visit of LA38-0411 being Visit 1 of LA38-EXT. Patients who had been treated with deferiprone during LA38-0411 continued to receive deferiprone for up to 2 years (Group 1), while those who had been treated with deferoxamine were switched to deferiprone for treatment up to 2 years (Group 2) in LA38-EXT. The dosage of deferiprone was 25–33 mg/kg three times a day (t.i.d.).

#### 4 STUDY PROCEDURES

The procedures and assessments to be conducted at each study visit are shown in Table 1.

Statistical Analysis Plan LA38-EXT

Table 1 Table of study procedures

ApoPharma Inc.

| | | | | | | | | | | Vioit 0 |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Visit 1 | Blood<br>Draws <sup>2</sup> | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | or Early<br>Termination |
| Week: | 0 | | 13 | 26 | 39 | 52 | 65 | 78 | 91 | 104 |
| Informed consent/assent | × | | | | | | | | = = = | |
| Eligibility criteria | X | | | | | | | | | |
| Prior and concomitant medications | × | | × | × | × | × | × | × | × | × |
| Transfusion information (if applicable) <sup>3</sup> | X | × | × | × | × | × | × | × | × | × |
| Serum pregnancy testing (if applicable) 4 | X | | × | × | × | × | × | × | × | × |
| Physical examination | X | | | | | × | | | | × |
| Vital signs (including weight and height) 5 | × | | × | × | × | × | × | × | × | × |
| 12-lead ECG | X | | | | | × | | | | × |
| Contraceptive counseling | X | | × | × | × | × | × | × | × | × |
| Serology | × | | | | | | | | | × |
| Hematology | × | × | X | X | × | × | × | × | × | × |
| Biochemistry 6 | × | | | X | | × | | × | | × |
| Serum ferritin | × | | × | × | X | X | X | × | × | × |
| Urinalysis | × | | | | | X | | | | × |
| Liver MRI | × | | | | | × | | | | × |
| Cardiac MRI T2* | × | | | | 12<br>1 | × | | | | × |

Statistical Analysis Plan LA38-EXT

ApoPharma Inc.

| Procedure | Visit 1 | Blood<br>Draws <sup>2</sup> | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9<br>or Early<br>Termination |
|---|---|---|---|---|---|---|---|---|---|---|
| Week: | 0 | | 13 | 26 | 39 | 52 | 65 | 78 | 91 | 104 |
| Dose calculation/verify and adjust dose level | × | | X | × | X | × | X | × | × | 12 |
| Collect used and unused study medication | | | X | X | X | X | X | × | × | × |
| Dispense study<br>medication | X | | X | X | × | X | X | × | × | |
| Dispense patient diary card | X | | X | X | X | X | X | × | X | |
| Review and collect<br>diary card | | | X | X | X | X | × | X | × | × |
| Adverse events | X | | X | X | X | X | X | × | × | × |

- 0411, the measures obtained at the baseline visit of the LA38-0411 study will be used as the baseline measures for LA38-EXT as well.) deferoxamine in LA38-0411 and will now be receiving deferiprone for the first time. (For patients who received deferiprone in LA38-Visit 1 of study LA38-EXT is also the final visit of study LA38-0411. It serves as the baseline visit for those patients who received
- For Group 1, hematology testing is to be done monthly throughout the study. For Group 2, it is to be done weekly up to Visit 3 (Week 26), biweekly up to Visit 5 (Week 52), and monthly thereafter. At the quarterly site visits, this testing will be done as part of the routine procedures, and at the other time points it can be done at a local laboratory instead of at the site.
- Record volume of blood that the patient received during the transfusion, and the mean hematocrit of the packed red blood cell units transfused m
- 5 Females of childbearing potential only
- Height will be measured only at Visits 1, 5, and 9
- <sup>6</sup> At Visits 1, 3, 5, 7, and 9, the blood sample must be drawn following a 10-hour fast

# 4.1 Method of Assignment to Treatment

Not applicable. All patients in this extension study received deferiprone.

### 4.2 Blinding Procedures

Not applicable.

#### 4.3 Allocation of Patient Numbers

All patients in LA38-0411 were assigned a unique 6-digit number, where the first 3 digits represent the site code and the last 3 were sequentially assigned to each patient who signed the ICF. These assigned numbers were maintained when patients continued on to this extension study of LA38-EXT.

### 4.4 Treatment Compliance

Compliance reported in the eCRF was based on the patient's diary and on the return of used and unused medication containers. If compliance was greater than 100% and the patient reported taking all doses as prescribed, compliance would be reported as 100% in the eCRF. Under-compliance < 80% and over-compliance >120% were to be reported as a protocol deviation, unless under-compliance was due to treatment interruption because of infection or neutropenia or other extenuating circumstances.

### 5 MEASUREMENTS AND EVALUATIONS

### 5.1 Efficacy Measurements

#### 5.1.1 Liver Iron Concentration

MRI scans for liver iron were performed at Visit 1, Visit 5, and Visit 9 (or early termination).

#### 5.1.2 Cardiac MRI T2\*

MRI scans for the assessment of cardiac MRI T2\* were performed at Visit 1, Visit 5, and Visit 9 (or early termination).

#### 5.1.3 Serum Ferritin

Serum ferritin was assessed at the start of the extension study and quarterly thereafter.

### **5.2** Safety Measurements

#### **5.2.1** Adverse Events

An adverse event (AE) is any untoward medical occurrence in a patient who is administered a pharmaceutical or other therapeutic product in a clinical study, not necessarily having a causal relationship with the product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a product, whether or not considered related to that product.

#### **5.2.2** Serious Adverse Events

An SAE is an adverse event occurring at any dose that results in any of the following outcomes:

- Death
- A life-threatening adverse event
- Inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant disability or incapacity
- A congenital anomaly in the offspring of a patient who received the study treatment
- An important adverse event that does not result in death, is not life-threatening, and does not necessitate hospitalization but which in the investigator's judgment may jeopardize the patient and may necessitate medical or surgical intervention to prevent one of those outcomes. Examples include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or treatment-related substance abuse.

# 5.2.3 Adverse Events of Special Interest

### 5.2.3.1 Neutropenia

Patients taking deferiprone were monitored for neutropenia, defined as a confirmed absolute neutrophil count (ANC) less than  $1.5 \times 10^9$ /L. Categories of neutropenia are as follows:

• Mild: A confirmed ANC  $< 1.5 \times 10^9/L$  but  $\ge 1.0 \times 10^9/L$ 

• Moderate: A confirmed ANC < 1.0 x  $10^9/L$  but  $\ge 0.5$  x  $10^9/L$ 

• Severe: A confirmed ANC  $< 0.5 \times 10^9$ /L. Severe neutropenia is also

referred to as agranulocytosis.

For a case of neutropenia to be confirmed, there must be 2 consecutive counts, a maximum of 3 days apart, that are both less than the specified value. If both counts are below 1.5 x  $10^9/\text{L}$  but are not in the same severity category, a third count was required to determine the severity.

#### 5.2.3.2 Infections

If the patient developed fever or any type of infection during the study, deferiprone was to be interrupted immediately and neutrophil count should be obtained and monitored more frequently (every 2 days if ANC  $<1.5 \times 10^9$ /L). Patients should be advised to report immediately to their physician any symptoms indicative of infection such as fever, sore throat, and flu-like symptoms. Patients has been provided with an emergency services card with contact information, and the patient/legal guardian will be advised to carry this card at all times. In presence of confirmed fever and/or infection, they would be required to have their neutrophil counts tested as soon as possible and no later than 24 hours after the symptoms of infection was detected. Therapy with deferiprone could be re-initiated once all symptoms had been resolved and it was deemed safe by the investigator.

### 5.2.4 Laboratory Measurements

The following laboratory tests had been performed:

- **Hematology** (for Group 1, monthly throughout the study; for Group 2, weekly for the first 6 months, biweekly for the next 6 months, and monthly thereafter): hemoglobin, total WBC count, ANC, and platelet count
- **Biochemistry** (semi-annually; Visits 1, 3, 5, 7, and 9): total protein, GGT, lactate dehydrogenase (LDH), sodium, potassium, chloride, fasting glucose, total and direct bilirubin (indirect bilirubin will be calculated by the sponsor), AST, ALT, albumin, blood urea nitrogen, calcium, creatinine, uric acid, alkaline phosphatase, and amylase
- Serology (Visits 1 and 9): Hepatitis B and C and HIV testing
- Urinalysis (annually; Visits 1, 5, and 9): pH, specific gravity, glucose, protein, ketones, blood, and (if indicated by the dipstick results), sediment microscopy. If there is blood in the urine or three or more "plus signs" for protein, samples must be sent for microscopy.
- Pregnancy (quarterly; Visits 1–9): serum pregnancy test

### **5.2.5** Other Safety Measurements

### 5.2.5.1 Physical Examination

At Visits 1, 5, and 9, the investigator or a qualified delegate performed a physical examination of the following organs and systems: head, ears, eyes, nose, throat and neck, respiratory system, cardiovascular system, gastrointestinal system, musculoskeletal system, central and peripheral nervous system, skin, thyroid, and general constitution.

### 5.2.5.2 Vital Signs

Temperature, heart rate, respiration rate, and systolic and diastolic blood pressure were measured at each visit.

Weight was measured at each visit, and height was measured at Visits 1, 5, and 9.

# 5.2.5.3 Electrocardiogram

A standard 12-lead ECG was performed at Visits 1, 5, and 9. As a minimum, the following parameters had been assessed: HR, PR, QRS, QT, QTcF, QTcB. The results were interpreted by the investigator, and the overall interpretation had been documented.

#### 5.2.5.4 Concomitant Medications

Information about prior and concomitant medications was collected at each visit. The following was to be recorded in the source documents and eCRFs:

- Any medications that the patient continues to take during the trial
- Any medications that the patient starts to take during the trial

#### 6 STATISTICAL ANALYSIS

#### 6.1 Endpoints

#### 6.1.1 Primary Endpoints

- Adverse events (AEs): Frequency, severity, time to onset (the start date of AE minus the start date of exposure to treatment), duration (the stop date of AE minus the start date of AE), and relatedness to study product
- Serious adverse events (SAEs): Frequency and relatedness to study product
- Number of discontinuations due to AEs

### **6.1.2** Secondary Endpoints

The time points for the efficacy assessments are defined below. Since the baseline measures are by definition those taken prior to the start of deferiprone therapy, "baseline" is defined differently for the two groups, as follows:

- Group 1: For patients who received deferiprone in LA38-0411, the baseline visit of that study will be treated as the baseline visit of LA38-EXT as well. Thus, Week 0 of the extension study will be Year 1 (i.e., the completion of one year of deferiprone treatment), Week 52 will be Year 2, and Week 104 will be Year 3 of deferiprone treatment.
- Group 2: For patients who received deferoxamine in LA38-0411, the start of the extension study (Week 0) will be treated as the baseline visit. For this group, therefore, Week 52 will be Year 1, and Week 104 will be Year 2 of deferiprone treatment.

Efficacy endpoints for deferiprone therapy are provided below. For Group 1, the change from baseline to Year 1 is derived from study LA38-0411. For Group 2, there is no Year 3 of deferiprone treatment.

- The change from baseline to Year 1 (both groups; Group 1 data are from LA38-0411), from baseline to Year 2 (both groups), and from baseline to Year 3 (Group 1 only) in liver iron concentration (LIC), as measured by magnetic resonance imaging (MRI)
- The change from baseline to Year 1 (both groups; Group 1 data are from LA38-0411), from baseline to Year 2 (both groups), and from baseline to Year 3 (Group 1 only) in cardiac MRI T2\*
- The change from baseline to Year 1 (both groups; Group 1 data are from LA38-0411 data), from baseline to Year 2 (both groups), and from baseline to Year 3 (Group 1 only) in serum ferritin
- Responder analysis, defined as the percentage of patients who show a ≥20% decline from baseline in LIC or serum ferritin or a ≥20% increase from baseline in cardiac MRI T2\* at Year 1 (both groups; Group 1 data are from LA38-0411), at Year 2 (both groups), and at Year 3 (Group 1 only)

In addition to the above analyses, the change from baseline to end of LA38-041 for deferoxamine and the change from baseline to end of LA38-EXT for deferiprone in Group 2 will be compared. The purpose of this analysis is to assess if deferiprone could maintain or even further improve LIC and MRI T2\* after the patients were switched therapy.

# **6.2** Study Populations

Study populations intended for analysis are defined as follows: Intent-to-Treat (ITT), Per-Protocol (PP), and Safety. The ITT population will represent the primary analysis population to evaluate all efficacy endpoints. The efficacy endpoints will also be analyzed for the PP population, which is the secondary analysis population.

# **6.2.1** Intent-to-Treat Population

The ITT population will include all randomized patients who received at least one dose of study drug and have a baseline and at least one post-baseline efficacy assessment.

# 6.2.2 Per Protocol Population

The Per-Protocol (PP) population will include all enrolled patients who complete the study, have no major protocol violations, and have an efficacy assessment at the end of the study. Prior to database lock, patients with major protocol violations will be reviewed and excluded, where appropriate, from the PP population. Major protocol violations will include (but not be limited to) the following:

- Patients who were not compliant with the treatment (<80% compliance)
- Patients who took iron chelator medications other than the assigned study medication during the course of the study

### 6.2.3 Safety Population

The safety population will include all enrolled patients who took at least one dose of study drug.

#### 6.3 Data Analysis

### 6.3.1 Patient Disposition and Drug Exposure

Patient disposition will be summarized and presented, including the number and percentages of patients who were enrolled, received at least one dose of study medication, completed the study, and withdrew (including reasons for withdrawals). For each patient, the number of doses taken will be computed from the study drug dispensing and accountability eCRFs obtained at each visit. The overall mean of total daily dose taken during the study will be summarized with descriptive statistics.

#### **6.3.2** Patient Characteristics

Baseline characteristics for continuous variables will be summarized with descriptive statistics such as mean, standard deviation, minimum, median and maximum values. Baseline characteristics for discrete variables will be summarized with frequency tables.

### 6.3.3 Analysis of Efficacy

Changes in LIC, in cardiac MRI T2\*, and in serum ferritin from baseline to Year 1 (both groups; Group 1 data are from LA38-0411), from baseline to Year 2 (both groups), and from

baseline to Year 3 (Group 1 only) will be summarized with descriptive statistics and will be tested against no change using a one-sample t-test. The changes in these 3 efficacy measures from the start of deferiprone therapy to the last visit of LA38-EXT in all patients, irrespective of whether deferiprone therapy was initiated in LA38-0411 or in LA38-EXT, will also be tested using a one-sample t-test. In addition, the percentages of responders will be tabulated for Year 1 (both groups; Group 1 data are from LA38-0411), for Year 2 (both groups), and for Year 3 (Group 1 only) of deferiprone therapy. The change from baseline to end of LA38-041 for deferoxamine and the change from baseline to end of LA38-EXT for deferiprone in Group 2 will be compared.

#### 6.3.4 Analysis of Safety

The incidences of AEs and SAEs reported from the start of deferiprone therapy for all patients will be tabulated. For patients continuing on deferiprone, this time period will be from the start of LA38-0411 to the completion of LA38-EXT; for those switching to deferiprone, it will be from the start of LA38-EXT to the completion of LA38-EXT. AEs will be summarized by worst severity and by relationship to the study medication. Time to onset and duration of all SAEs, of AEs of special interest such as neutropenia, agranulocytosis, increased ALT, and arthralgia: 1) the mean time to the first onset and the mean time to the last recurrence will be calculated, and 2) the mean duration for the first episode and the mean duration for any recurrent episodes, excluding the first episode, will be calculated for all SAEs and AEs of special interest.

The percentage of discontinuations due to AEs will be calculated, and the AEs leading to discontinuation will be summarized in a frequency table.

Laboratory data (hematology and chemistry) will be summarized using descriptive statistics for continuous variables and frequency tables for discrete variables. The incidences of out-of-range data will be tabulated, and the changes from baseline to the end of study will be presented in shift tables.

#### 14 SUMMARY TABLES AND FIGURES

Note: The final numberings for tables and/or figures in the clinical study report can be changed if more tables and/or figures are added in addition to those in the SAP.

#### **TABLES**

#### 14.1 Disposition, Demographics and Baseline Data

- Table 14.1.1 Patient disposition
- Table 14.1.2 Number of patients in the ITT, PP, and safety populations
- Table 14.1.3 Number of patients by study site
- Table 14.1.4 Reasons for not completing the study
- Table 14.1.5 Demographics data
- Table 14.1.6 LIC, cardiac MRI T2\*, serum ferritin at baseline
- Table 14.1.7 Medical history
- Table 14.1.8 Vital signs at baseline
- Table 14.1.9 Weight and height at baseline

#### 14.2 Efficacy Analyses

#### 14.2.1 LIC

- Table 14.2.1.1 LIC at each assessment
- Table 14.2.1.2 Change in LIC at each follow-up assessment
- Table 14.2.1.3 Change in LIC for DFO+DFP group Data from the extension study
- Table 14.2.1.4 Change in LIC for DFO and DFO+DFP group
- Table 14.2.1.5 Responder analysis in LIC defined as ≥ 20% decline in LIC from baseline
- Table 14.2.1.6 Responder analysis in LIC defined as ≥ 20% decline in LIC from baseline for
- DFO+DFP group Data from the extension study

#### 14.2.2 Cardiac MRI T2\*

- Table 14.2.2.1 Cardiac MRI T2\* at each assessment
- Table 14.2.2.2 Change cardiac MRI T2\* at each follow-up assessment
- Table 14.2.2.3 Change in cardiac MRI T2\* for DFO+DFP group Data from the extension Study
- Table 14.2.2.4 Change in cardiac MRI T2\* for DFO and DFO+DFP group
- Table 14.2.2.5 Responder analysis in cardiac MRI T2\* defined as  $\geq$  20% increase in cardiac MRI T2\* from baseline

Table 14.2.2.6 Responder analysis in cardiac MRI T2\* defined as  $\geq$  20% increase in cardiac MRI T2\* baseline for DFO+DFP group – Data from the extension study

#### 14.2.3 Serum Ferritin

Table 14.2.3.1 Serum ferritin at each assessment

Table 14.2.3.2 Change in serum ferritin at each follow-up assessment

Table 14.2.3.3 Change in serum ferritin for DFO+DFP group – Data from the extension study

Table 14.2.3.4 Responder analysis in serum ferritin defined as  $\geq$  20% decline in serum ferritin from baseline

Table 14.2.3.5 Responder analysis in serum ferritin defined as  $\geq$  20% decline in serum ferritin from baseline for DFO+DFP group – Data from the extension study

#### 14.3 Safety Analyses

#### 14.3.1 Adverse Events

Table 14.3.1.1 Overall summary of adverse events – Safety population

Table 14.3.1.2 Summary of adverse events – Safety population

Table 14.3.1.3 Summary of most common adverse events (≥5% in total) – Safey population

Table 14.3.1.4 Summary of adverse drug reactions – Safety population

Table 14.3.1.5 Summary of most common adverse drug reactions (≥5% in total) – Safety population

Table 14.3.1.6 Summary of serious adverse events – Safety population

Table 14.3.1.7 Summary of serious adverse drug reactions – Safety population

Table 14.3.1.8 Summary of adverse events by causality – Safety population

Table 14.3.1.9 Time to the first onset of SAEs – Safety population

Table 14.3.1.10 Time to the first onset of AEs of special interest such as neutropenia, agranulocytosis, increased ALT, arthralgia – Safety population

Table 14.3.1.11 Time to the last recurrence of SAEs – Safety population

Table 14.3.1.12 Time to the last recurrence of AEs of special interest such as neutropenia, agranulocytosis, increased ALT, arthralgia – Safety population

Table 14.3.1.13 Duration of the first onset of SAEs – Safety population

Table 14.3.1.14 Duration of the first onset of AEs of special interest such as neutropenia, agranulocytosis, increased ALT, arthralgia – Safety population

Table 14.3.1.15 Duration of the last recurrence of SAEs – Safety population

Table 14.3.1.16 Duration of the last recurrence of AEs of special interest such as neutropenia, agranulocytosis, increased ALT, arthralgia – Safety population

### 14.3.2 Vital Signs

Table 14.3.2.1 Temperature at each assessment – Safety population

Table 14.3.2.2 Change in temperature from baseline to each follow-up assessment – Safety population

Note: Similar tables will be produced for resting heart rate, respiration, systolic blood pressure, and diastolic blood pressure.

#### 14.3.3 Weight and Height

Table 14.3.3.1 Weight at each assessment – Safety population

Table 14.3.3.2 Change in weight from baseline to last assessment – Safety population

Table 14.3.3.1 Height at each assessment – Safety population

Table 14.3.3.2 Change in height from baseline to last assessment – Safety population

#### 14.3.4 Concomitant Medications

Table 14.3.4.1 Concomitant medications – Safety population

#### 14.3.5 12-Lead ECG

Table 14.3.5.1 Heart rate of 12-Lead ECG at each assessment – Safety population Table 14.3.5.2 Change in heart rate of 12-Lead ECG from baseline to each follow-up assessment – Safety population

Note: Similar tables will be produced for PR, QRS, QT, QTcF, and QTcB.

Table 14.3.5.3 Shift table for clinically significant abnormality for 12-Lead ECG – Safety population

### 14.3.6 Laboratory Data

#### 14.3.6.1 Hematology

Table 14.3.6.1.1 Hemoglobin at each assessment – Safety population

Table 14.3.6.1.2 Change in hemoglobin from baseline to each follow-up assessment – Safety population

Table 14.3.6.1.3 Shift table for hemoglobin in abnormal range at baseline vs. last assessment – Safety population

Note: Similar tables will be produced for total white blood cell (WBC), absolute neutrophil count (ANC), and platelets.

### 14.3.6.2 Biochemistry

Table 14.3.6.2.1 Total protein at each assessment – Safety population

Table 14.3.6.2.2 Change in total protein from baseline to each follow-up assessment – Safety population

Table 14.3.6.2.3 Shift table for total protein in abnormal range at baseline vs. last assessment – Safety population

Note: Similar tables will be produced for GGT, lactate dehydrogenase (LDH), sodium, potassium, chloride, glucose (fasting at screening visit only), total, direct and indirect bilirubin, AST, ALT, albumin; blood urea nitrogen, calcium, creatinine, uric acid, alkaline phosphatase, and amylase.

### 14.3.6.3 Serology

Table 14.3.6.3.1 HIV at each assessment – Safety population Note: Similar tables will be produce for Hepatitis B and C. – Safety population

# 14.3.7 Pregnancy test

Table 14.3.7.1 Female patients with positive pregnancy test during the study – Safety population

### 14.4 Treatment compliance

14.4.1 The number and percent of patients who had compliance <80% or >120% during the study – Safety population

#### 14.5 Transfusion information

Table 14.5.1 Overall mean of transfusional iron input (mg/kg/day) during the study – Safety population

# 14.6 Total daily dose

Table 14.6.1 Overall mean of total daily dose (mg/kg/day) during the study – Safety population

#### **FIGURES**

### 14.2 Efficacy

Figure 14.2.1 Mean line graph for LIC over time – ITT population

Figure 14.2.2 Mean line graph for cardiac MRI T2\* over time – ITT population

Figure 14.2.3 Mean line graph for serum ferritin over time – ITT population

Figure 14.2.4 Mean line graph for the change in LIC from baseline to the end of study – ITT population

Figure 14.2.5 Mean line graph for the change in cardiac MRI T2\* from baseline to the end of study – ITT population

Figure 14.2.6 Mean line graph for the change in serum ferritin from baseline to the end of study – ITT population

### 14.3 Safety

#### 14.3.1 Hematology

Figure 14.3.1.1 Mean line graph for hemoglobin over visit – Safety population Figure 14.3.1.2 Proportion of patients with abnormal hemoglobin at each assessment – Safety population

Note: Similar graphs will be produced for total white blood cell (WBC), absolute neutrophil count (ANC), and platelets.

#### 14.3.2 Biochemistry

Figure 14.3.2.1 Mean line graph for total protein over visit – Safety population Figure 14.3.2.2 Proportion of patients with abnormal total protein at each assessment – Safety population

Note: Similar tables will be produced for GGT, lactate dehydrogenase (LDH), sodium, potassium, chloride, glucose (fasting at screening visit only), total, direct and indirect bilirubin, AST, ALT, albumin; blood urea nitrogen, calcium, creatinine, uric acid, alkaline phosphatase, and amylase.

#### 16 DATA LISTINGS

Note: The final numberings for patient data listings in the clinical study report can be changed if more patient data listings are made in the addition to those in the SAP.

### 16.2 Patient Data Listings

- 16.2.1 Listing of informed consent
- 16.2.2 Listing of demographics
- 16.2.3 Listing of primary diagnosis
- 16.2.4 Listing of transfusion history
- 16.2.5 Listing of vital signs including height, weight
- 16.2.6 Listing of physical examination
- 16.2.7 Listing of 12-lead electrocardiogram
- 16.2.8 Listing of urinalysis
- 16.2.9 Listing of hematology
- 16.2.10 Listing of LIC
- 16.2.11 Listing of cardiac MRI T2\*
- 16.2.12 Listing of chemistry
- 16.2.13 Listing of serology
- 16.2.14 Listing of pregnancy
- 16.2.15 Listing of urine microscopy
- 16.2.16 Listing of serum ferritin
- 16.2.17 Listing of dose verification
- 16.2.18 Listing of disposition
- 16.2.19 Listing of compliance
- 16.2.20 Listing of medical history
- 16.2.21 Listing of medication
- 16.2.22 Listing of medical events
- 16.2.23 Listing of adverse events
- 16.2.24 Listing of exposure
- 16.2.25 Listing of local labs
- 16.2.26 Listing of transfusion information
- 16.2.27 Listing of SAEs
- 16.2.28 Listing of withdrawals due to AEs

#### 17 TABLE SHELLS

The following table shells provide a framework for the display of data from this study. These tables may not be produced exactly as shown in the shells, but are intended to reflect the general layout of the data that will be included in the clinical study report.

Note that 'c' in the table shells indicates an alphanumeric character and 'x' indicates a number from 0 to 9.

If the same data points are collected at more than one visit, the results will be summarized in Table x.x for baseline, x.x-1 for visit 1, x.x-2 for visit 2 and so on.

Table 14.1.1 Patient disposition

| | Treati | ment |
|------------|-----------|-----------|
| | DFP+ DFP | DFO+DFP |
| Enrolled | Xxx | xxx |
| Exposed* | xxx (xx%) | xxx (xx%) |
| Completed* | xxx (xx%) | xxx (xx%) |
| Withdrawn* | xxx (xx%) | xxx (xx%) |

Data source: 16.2.18 Listing of disposition

Note: \*Percentages are based on the number of enrolled patients in each treatment group.

Table 14.1.2 Number of patients in the ITT, PP, and safety populations

| | | Trea | tment |
|-------------------|-----------------|---------|---------|
| | | DFP+DFP | DFO+DFP |
| _ | LIC | xxx | xxx |
| ITT population | Cardiac MRI T2* | xxx | xxx |
| = | Serum Ferritin | xxx | xxx |
| | LIC | xxx | xxx |
| PP population | Cardiac MRI T2* | xxx | xxx |
| | Serum Ferritin | xxx | xxx |
| Safety population | | xxx | xxx |

Data source: 16.2.10 Listing of LIC, 16.2.11 Listing of cardiac MRI T2\*, and 16.2.16 Listing of serum ferritin, and 16.2.24 Listing of exposure

1.45

Table 14.1.3 Number of patients by study site

| | Tre | atment |
|------------|---------|---------|
| Study Site | DFP+DFP | DFO+DFP |
| 001 | xxx | xxx |
| 002 | XXX | xxx |
| *** | ••• | ••• |
| Total | xxx | XXX |

Data source: 16.2.2 Listing of demographics

Table 14.1.4 Reasons for not completing the study

| | | Trea | tment |
|-----------------------|--------|----------|----------|
| | | DFP+DFP | DFO+DFP |
| N (%) | | xx (100) | xx (100) |
| Reason | Detail | | |
| Adverse event | Ccccc | xx (xx) | xx (xx) |
| 1 tavoise event | Ccccc | xx (xx) | xx (xx) |
| Voluntary | Ccccc | xx (xx) | xx (xx) |
| withdrawal | Ccccc | xx (xx) | xx (xx) |
| Lost to follow-up | Ccccc | xx (xx) | xx (xx) |
| 2000 to follow up | Ccccc | xx (xx) | xx (xx) |
| Investigator decision | Ccccc | xx (xx) | xx (xx) |
| mivestigated decision | Ccccc | xx (xx) | xx (xx) |
| Protocol violation | Ccccc | xx (xx) | xx (xx) |
| 1 Totogor Violation | Ccccc | xx (xx) | xx (xx) |
| Other | Ccccc | xx (xx) | xx (xx) |
| | Ccccc | xx (xx) | xx (xx) |
| Total | | xx (xx) | xx (xx) |

Data source: 16.2.18 Listing of disposition

Table 14.1.5 Demographics data

| | Treat | ment | |
|---|---|---|---|
| | DFP+DFP | DFO+DFP | |
| N | Xxx | XXX | p-value§ |
| Age (years): | | | 0.xxxx |
| Mean ± SD | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| (Min, Median, Max) | (xx.x, xx.x, xx.x) | (xx.x, xx.x, xx.x) | |
| Sex: n (%) | | | 0.xxxx |
| Female | xx (xx) | xx (xx) | |
| Male | xx (xx) | xx (xx) | |
| Ethnic Origin: n (%) | | | 0.xxxx |
| Hispanic/Latino | xx (xx) | xx (xx) | |
| Other | xx (xx) | xx (xx) | |
| Racial Origin: n (%) | | | 0.xxxx |
| White | xx (xx) | xx (xx) | |
| Black | xx (xx) | xx (xx) | |
| Asian | xx (xx) | xx (xx) | |
| Native American | xx (xx) | xx (xx) | |
| Native Hawaiian/Other Pacific Islander | xx (xx) | xx (xx) | |
| Multi-Racial | xx (xx) | xx (xx) | |

§ T-test for age; Fisher's exact test for sex, ethnic origin, and racial origin

Data source: 16.2.2 Listing of demographics

Table 14.1.6 LIC, cardiac MRI T2\*, and serum ferritin at baseline

| | Tre | atment | |
|---|---|---|---|
| | DFP+DFP | DFO+DFP | |
| N | xxx | xxx | |
| | Mean ± SD | Mean ± SD | P-value (t-test) |
| | (Min, Max) | (Min, Max) | 1 - varue (t-test) |
| LIC (mg/g dw) | xx.x ± xx.x<br>(xx.x, xx.x) | $xx.x \pm xx.x$<br>(xx.x, xx.x) | 0.xxxx |
| Cardiac MRI T2* | xx.x ± xx.x | XX.X ± XX.X | 0.xxxx |
| (ms) | (xx.x, x.xx) | (xx.x, xx.x) | |
| Serum Ferritin | xxxx ± xxxx | xxxx ± xxxx | 0.xxxx |
| (µg/L) | (xxxx, xxxx) | (xxxx, xxxx) | |

Data source: 16.2.10 Listing of LIC, 16.2.11 Listing of cardiac MRI T2\*, 16.2.16 Listing of serum ferritin

Table 14.1.7 Medical history

| | | Treatment | | |
|---|---|---|---|---|
| | DFP- | +DFP | DFO | +DFP |
| N | X | XXX | | xx |
| Illness/Event by MedDRA Primary System Organ Class and Preferred Term | Resolved Ongoing n (%) n (%) | | Resolved<br>n (%) | Ongoing n (%) |
| Сссссс | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Сссссс | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| ccccc | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| ссссс | xx (xx) | xx (xx) | xx (xx) | xx (xx) |

Data source: 16.2.20 Listing of medical history

Table 14.1.8 Vital signs at baseline

| | Treatment | | |
|---|---|---|---|
| | DFP+DFP | DFO+DFP | |
| N | xxx | xxx | |
| Vital Sign: | Mean ± SD<br>(Min, Max) | Mean ± SD<br>(Min, Max) | P-value (T-test) |
| Temperature (°C) | $xx.x \pm xx.x$ $(xx, xx)$ | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Resting Heart Rate (/min) | xxx.x ± xxx.x<br>(xxx, xxx) | xxx.x ± xxx.x<br>(xxx, xxx) | 0.xxxx |
| Respiration (/min) | $xx.x \pm xx.x$<br>(xx, xx) | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Systolic Blood Pressure (mmHg) | xxx.x ± xxx.x<br>(xxx, xxx) | xxx.x ± xxx.x<br>(xxx, xxx) | 0.xxxx |
| Diastolic Blood<br>Pressure (mmHg) | xxx.x ± xxx.x<br>(xxx, xxx) | xxx.x ± xxx.x<br>(xxx, xxx) | 0.xxxx |

Data source: 16.2.5 Listing of vital signs including height and weight

Table 14.1.9 Weight and height at baseline

| | Treat | | |
|---|---|---|---|
| | DFP+DFP | DFO+DFP | |
| N | xxx | xxx | |
| | Mean ± SD<br>(Min, Max) | Mean ± SD<br>(Min, Max) | P-value (T-test) |
| Weight (kg) | $xx.x \pm xx.x$<br>(xx, xx) | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Height (cm) | $xxx.x \pm xxx.x$<br>(xxx, xxx) | $xxx.x \pm xxx.x$<br>(xxx, xxx) | 0.xxxx |

§For patients who had separate screening and baseline visits, height was measured only at screening Data source: 16.2.5 Listing of vital signs including height and weight

Table 14.2.1.1 LIC at each assessment

| | | Trea | atment | |
|---------------|-----------|-----------------|-----------------|----------|
| | | DFP+DFP | DFO+DFP | |
| | Visit | N | N | P-value |
| | | Mean ± SD | Mean ± SD | (T-test) |
| | | (Min, Max) | (Min, Max) | |
| | Baseline | xxx | xxx | 0.xxxx |
| | Buschine | xx.x ± xx.x | $xx.x \pm xx.x$ | • |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 6 | xxx | xxx | 0.xxxx |
| | 1,10,11,1 | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Year 1 | xxx | xxx | 0.xxxx |
| LIC (mg/g dw) | | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Year 2 | xxx | xxx | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Year 3 | xxx | xxx | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |

Data source: 16.2.10 Listing of LIC

Table 14.2.1.2 Change in LIC at each follow-up assessment

| | | Treatment | | |
|---------------|---------|-----------------|-----------------|----------|
| | | DFP+DFP | DFO+DFP | |
| | Visit | N | N | P-value |
| | | Mean ± SD | Mean ± SD | (T-test) |
| | | (Min, Max) | (Min, Max) | |
| | Month 6 | xxx | xxx | 0.xxxx |
| | Wiolidi | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Year 1 | xxx | xxx | 0.xxxx |
| | 1 Cal 1 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| Change in LIC | | (xx.x, xx.x) | (xx.x, xx.x) | |
| (mg/g dw) | Year 2 | xxx | xxx | 0.xxxx |
| | Teal 2 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Year 3 | xxx | xxx | 0.xxxx |
| | 10013 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |

Data source: 16.2.10 Listing of LIC

Table 14.2.1.3 Change in LIC for DFO+DFP group - Data from the extension study

| | | DFO+DFP | |
|---|---|---|---|
| | Visit | N<br>Mean ± SD<br>(Min, Max) | P-value<br>(One sample T-test) |
| From Year 1 t Year 2 | Year 1 to | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | 0.xxxx |
| (mg/g dw) | From<br>Year 1 to<br>Year 3 | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | 0.xxxx |

Data source: 16.2.10 Listing of LIC

Table 14.2.1.4 Change in LIC for DFO and DFO+DFP groups

| | | Trea | Treatment | |
|---------------|--------|-----------------|-----------------|----------|
| | | DFO* | DFO+DFP* | |
| | Visit | N | N | P-value |
| | | Mean ± SD | Mean ± SD | (T-test) |
| | | (Min, Max) | (Min, Max) | |
| Change in LIC | End of | xxx | Xxx | 0.xxxx |
| (mg/g dw) | Study | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| (mg/g dw) | Study | (xx.x, xx.x) | (xx.x, xx.x) | |

Data source: 16.2.10 Listing of LIC

Note: \*Patients in DFO come from LA38-0411 and patients in DFO+DFP comes from LA38-EXT.

Table 14.2.1.5 Responder analysis in LIC defined as ≥ 20% decline in LIC from baseline.

| | | Treatmer | | | |
|---|---|---|---|---|---|
| | DFP+ | -DFP | DFO+DI | P | P-value<br>(Fisher's exact test) |
| | N | n (%) | N | n (%) | 0.xxxx |
| Year 1 | xxx | xx (xx%) | xxx | xx (xx%) | 0.xxxx |
| Year 2 | xxx | xx (xx%) | xxx | xx (xx%) | 0.xxxx |
| Year 3 | xxx | xx (xx%) | xxx | xx (xx%) | 0.xxxx |

Data source: 16.2.10 Listing of LIC

Table 14.2.1.6 Responder analysis in LIC defined as  $\geq$  20% decline in LIC from baseline for DFO+DFP group – Data from the extension study.

| | Treatment | |
|--------|-----------|----------|
| | DFO+DFP | |
| | N | n (%) |
| Year 1 | xxx | xx (xx%) |
| Year 2 | xxx | xx (xx%) |

Data source: 16.2.10 Listing of LIC

Table 14.2.2.1 Cardiac MRI T2\* at each assessment

| | | Trea | tment | |
|--------------|----------|-----------------|-----------------|----------|
| | | DFP+DFP | DFO+DFP | |
| | Visit | N | N | P-value |
| | | Mean ± SD | Mean ± SD | (T-test) |
| | | (Min, Max) | (Min, Max) | |
| | Baseline | xxx | xxx | 0.xxxx |
| | Dascille | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | • |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 6 | xxx | xxx | 0.xxxx |
| | Wionin o | $xx.x \pm xx.x$ | xx.x ± xx.x | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| Cardiac | Year 1 | xxx | xxx | 0.xxxx |
| | 1 Car 1 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| MRI T2* (ms) | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Year 2 | xxx | xxx | 0.xxxx |
| | Tour Z | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Year 3 | xxx | xxx | 0.xxxx |
| | Tour 5 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |

Data source: 16.2.11 Listing of cardiac MRI T2\*

Table 14.2.2.2 Change in cardiac MRI T2\* at each follow-up assessment

| | | Trea | | |
|-------------|--------------|-----------------|-----------------|----------|
| | | DFP+DFP | DFO+DFP | |
| | Visit | N | N | P-value |
| | | Mean ± SD | Mean ± SD | (T-test) |
| | | (Min, Max) | (Min, Max) | |
| | Month 6 | xxx | xxx | 0.xxxx |
| | I Trionian o | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Year 1 | xxx | xxx | 0.xxxx |
| Change in | 1000 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| cardiac MRI | | (xx.x, xx.x) | (xx.x, xx.x) | |
| T2* (ms) | Year 2 | xxx | xxx | 0.xxxx |
| 12 (1113) | 10412 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Year 3 | xxx | xxx | 0.xxxx |
| | | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |

Data source: 16.2.11 Listing of cardiac MRI T2\*

Table 14.2.2.3 Change in cardiac MRI T2\* for DFO+DFP group – Data from the extension study

| | | DFO+DFP | |
|---|---|---|---|
| | Visit | N<br>Mean ± SD<br>(Min, Max) | P-value<br>(One sample T-test) |
| Change in cardiac MRI | From<br>Year 1 to<br>Year 2 | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | 0.xxxx |
| T2* (ms) | From<br>Year 1 to<br>Year 3 | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | 0.xxxx |

Data source: 16.2.11 Listing of cardiac MRI T2\*

Table 14.2.2.4 Change in cardiac MRI T2\* for DFO and DFO+DFP groups

| 77 | 11 | Treatment | | |
|-------------------|--------|--------------|-----------------|----------|
| | | DFO* | DFO+DFP* | |
| | Visit | N | N | P-value |
| | | Mean ± SD | Mean ± SD | (T-test) |
| | | (Min, Max) | (Min, Max) | |
| Character conding | End of | xxx | Xxx | 0.xxxx |
| Change in cardiac | Study | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| MRI T2* (ms) | Study | (xx.x, xx.x) | (xx.x, xx.x) | |

Data source: 16.2.11 Listing of cardiac MRI T2\*

Note: \*Patients in DFO come from LA38-0411 and patients in DFO+DFP comes from LA38-EXT.

Table 14.2.2.5 Responder analysis in cardiac MRI T2\* defined as  $\geq$  20% increase in cardiac MRI T2\* from baseline.

| | Treatment | | | | |
|---|---|---|---|---|---|
| | DFP | DFP+DFP | | DFP | P-value<br>(Fisher's exact test) |
| | N | n (%) | N | n (%) | 0.xxxx |
| Year 1 | xxx | xx (xx%) | xxx | xx (xx%) | 0.xxxx |
| Year 2 | xxx | xx (xx%) | XXX | xx (xx%) | 0.xxxx |
| Year 3 | xxx | xx (xx%) | XXX | xx (xx%) | 0.xxxx |

Data source: 16.2.11 Listing of cardiac MRI T2\*

Table 14.2.2.6 Responder analysis in cardiac MRI T2\* defined as  $\geq$  20% increase in cardiac MRI T2\* from baseline for DFO+DFP group – Data from the extension study.

| | Treatment |
|------|-----------|
| DFO+ | DFP |
| N | n (%) |
| xxx | xx (xx%) |
| XXX | xx (xx%) |
| | DFO+ |

Data source: 16.2.11 Listing of cardiac MRI T2\*

Table 14.2.3.1 Serum ferritin each assessment

| | | Treatment | | |
|----------------|----------|-----------------|-----------------|----------|
| | | DFP+DFP | DFO+DFP | |
| | Visit | N | N | P-value |
| | | Mean ± SD | Mean ± SD | (T-test) |
| | | (Min, Max) | (Min, Max) | |
| | Baseline | xxx, | xxx | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 3 | xxx | xxx | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 6 | xxx | xxx | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 9 | xxx | xxx | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 12 | xxx | XXX | 0.xxxx |
| | | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 15 | xxx | xxx | 0.xxxx |
| | | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| Serum Ferritin | | (xx.x, xx.x) | (xx.x, xx.x) | |
| $(\mu g/L)$ | Month 18 | xxx | XXX | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 21 | xxx | xxx | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 24 | xxx | XXX | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 27 | xxx | XXX | 0.xxxx |
| | | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 30 | xxx | XXX | 0.xxxx |
| | | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 33 | xxx | xxx | 0.xxxx |
| | | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |

| | Treatment | | |
|---|---|---|---|
| | DFP+DFP | DFO+DFP | |
| Month 36 | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | 0.xxxx |

Data source: 16.2.16 Listing of serum ferritin

Table 14.2.3.2 Change in serum ferritin at each follow-up assessment

| | | Treatment | | |
|---|---|---|---|---|
| | | DFP+DFP | DFO+DFP | |
| | Visit | N | N | P-value |
| | | Mean ± SD | Mean ± SD | (T-test) |
| | | (Min, Max) | (Min, Max) | |
| | 26 4 2 | xxx | xxx | 0.xxxx |
| | Month 3 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 6 | xxx | xxx | 0.xxxx |
| _ = = _ = = | - Wolling | $-xx.x \pm xx.x$ | $xx.x \pm xx.x$ | = |
| Change in serum | | (xx.x, xx.x) | (xx.x, xx.x) | |
| ferritin (µg/L) | Month 9 | xxx | XXX | 0.xxxx |
| | | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 12 | xxx | XXX | 0.xxxx |
| | | xx.x ± xx.x | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 15 | xxx | XXX | 0.xxxx |
| | Wiolitii 13 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 18 | xxx | xxx | 0.xxxx |
| | IVIORUI 10 | $xx.x \pm xx.x$ | xx.x ± xx.x | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | = = = |
| | Month 21 | xxx | xxx | 0.xxxx |
| | Wionin 21 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Month 24 | xxx | xxx | 0.xxxx |
| | Wionui 24 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | (xx.x, xx.x) | |
| | | Treatment | | Essis a |
|---|---|---|---|---|
| | | DFP+DFP | DFO+DFP | él. |
| Month | 27 | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | 0.xxxx |
| Month | 30 | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | 0.xxxx |
| Month | 33 | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | 0.xxxx |
| Month | 36 | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | xxx<br>xx.x ± xx.x<br>(xx.x, xx.x) | 0.xxxx |

Data source: 16.2.16 Listing of serum ferritin

Table 14.2.3.3 Change in serum ferritin for DFO+DFP group – Data from the extension study

| | | DFO+DFP | |
|---|---|---|---|
| · | Visit | N | P-value |
| | | Mean ± SD | (One sample T-test) |
| | | (Min, Max) | |
| | From Month 12 | XXX | 0.xxxx |
| | to Month 15 | $xx.x \pm xx.x$ | |
| | 10 1101111 13 | (xx.x, xx.x) | |
| | From Month 12<br>to Month 18 | XXX | 0.xxxx |
| | | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | |
| | From Month 12<br>to Month 21 | XXX | 0.xxxx |
| Change in | | $xx.x \pm xx.x$ | |
| serum ferritin | | (xx.x, xx.x) | |
| (μg/L) | From Month 12 | XXX | 0.xxxx |
| (46,2) | to Month 24 | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | |
| | From Month 12 | XXX | 0.xxxx |
| | to Month 27 | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | |
| | From Month 12 | XXX | 0.xxxx |
| | to Month 30 | $xx.x \pm xx.x$ | |
| | | (xx.x, xx.x) | |

| | = 109 | DFO+DFP | |
|-------|---------------|-----------------|---------------------|
| - | Visit | N | P-value |
| | | Mean ± SD | (One sample T-test) |
| | | (Min, Max) | |
| | From Month 12 | xxx | 0.xxxx |
| | to Month 33 | $xx.x \pm xx.x$ | |
| == == | to Month 33 | (xx.x, xx.x) | |
| | From Month 12 | xxx | 0.xxxx |
| | to Month 36 | $xx.x \pm xx.x$ | |
| | to Month 20 | (xx.x, xx.x) | |

Data source: 16.2.16 Listing of serum ferritin

Table 14.2.3.4 Responder analysis in serum ferritin as defined ≥ 20% decline in serum ferritin from baseline.

| | | Treat | | | |
|---|---|---|---|---|---|
| | DFP | P+DFP DFO+DFP | | | P-value<br>(Fisher's exact test) |
| | N | n (%) | N | n (%) | 0.xxxx |
| Year 1 | xxx | xx (xx%) | xxx | xx (xx%) | 0.xxxx |
| Year 2 | xxx | xx (xx%) | XXX | xx (xx%) | 0.xxxx |
| Year 3 | xxx | xx (xx%) | xxx | xx (xx%) | 0.xxxx |

Data source: 16.2.16 Listing of serum ferritin

Table 14.2.3.5 Responder analysis in serum ferritin defined as  $\geq$  20% decline in serum ferritin from baseline for DFP+DFO group – Data from the extension study.

| | 7 | Treatment |
|--------|------|-----------|
| | DFO+ | DFP |
| | N | n (%) |
| Year 1 | xxx | xx (xx%) |
| Year 2 | xxx | xx (xx%) |

Data source: 16.2.16 Listing of serum ferritin

Table 14.3.1.1 Overall summary of adverse events

| | Trea | 50.6 | |
|---|---|---|---|
| | DFP+DFP | DFO+DFP** | |
| N | xxx | xxx | P-value<br>(Fisher's exact test) |
| Number of patients experiencing at least one AE | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patients experiencing at least one severe AE | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patients experiencing at least one serious AE | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patients experiencing at least one related* AE | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patient deaths | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patient withdrawals due to AEs | xx (xx%) | xx (xx%) | 0.xxxx |

<sup>\*</sup>Includes possibly, probably, and definitely related. Worst case scenario of causality between the investigator and company's assessment.

Data source: 16.2.23 Listing of adverse events

<sup>\*\*</sup>AEs occurred while on DFP treatment.

Table 14.3.1.2 Adverse events

| | Trea | | |
|---|---|---|---|
| | DFP+DFP | DFO+DFP | |
| | (N=xxx) | (N=xxx) | |
| | Exposure | Exposure | 1 |
| | (patient-years): x.xx | (patient-years):x.xx | |
| | Total Events: xxx | Total Events: xxx | 7 |
| System Organ Class<br>Preferred Term | n Patients (%) | n Patients (%) | P-value<br>(Fisher's<br>exact test) |
| CCCCCC | x (x.x) | x (x.x) | 0.xxxx |
| Ссссс | x (x.x) | x (x.x) | 0.xxxx |
| Ccccc | x (x.x) | x (x.x) | 0.xxxx |
| Ccccc | x (x.x) | x (x.x) | 0.xxxx |
| | | • | |

Note: Similar tables will be produced from Table 14.3.1.3 to Table 14.3.1.7

Data source: 16.2.23 Listing of adverse events

Table 14.3.1.8 Adverse events by causality

| | | Trea | tment |
|--------------------|---------------|--------------------|--------------------|
| | | DFP+DFP | DFO+DFP |
| | | (N=xxx) | (N=xxx) |
| System Organ Class | Relatedness | Patients reporting | Patients reporting |
| Preferred Term | (worst case) | (n=xx) | (n=xx) |
| CCCCCCC | | x (x.x) | x (x.x) |
| ccccc | Not Related* | x (x.x) | x (x.x) |
| | Related** | x (x.x) | x (x.x) |
| ccccc | Not Related | x (x.x) | x (x.x) |
| | Related* | x (x.x) | x (x.x) |
| ••••• | • • • • • • • | | • • • • • |

\*Not related

\*\*Possibly, Probably, or Definitely Related Data source: 16.2.23 Listing of adverse events Table 14.3.1.9 Time to the first onset of SAEs

| | | Treatment | | | |
|---|---|---|---|---|---|
| | | DFP+DFP | | DFO+DFP | |
| SAE | N | Mean ± SD (Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value<br>(T-test) |
| Ccccc | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Ccccc | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Ccccc | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |

Note: Similar table will be produced for Table 14.3.1.10.

Data source: 16.2.23 Listing of adverse events

Table 14.3.1.11 Time to the last recurrence of SAEs

| | | Treatment | | | |
|---|---|---|---|---|---|
| | | DFP+DFP | D | FO+DFP | = = |
| SAE | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value<br>(T-test) |
| Ccccc | xxx | $xx.x \pm xx.x$<br>(xx, xx) | Xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Ccccc | xxx | $xx.x \pm xx.x$<br>(xx, xx) | Xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| | xxx | $xx.x \pm xx.x$<br>(xx, xx) | Xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Ccccc | xxx | $xx.x \pm xx.x$<br>(xx, xx) | Xxx | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |

Note: Similar table will be produced for Table 14.3.1.12.

Data source: 16.2.23 Listing of adverse events

Table 14.3.1.13 Duration of the first onset of SAEs

| | | Treatment | | | |
|---|---|---|---|---|---|
| | | DFP+DFP | 1 | DFO+DFP | |
| SAE | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value<br>(T-test) |
| Ccccc | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Ссссс | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| • • • • | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Сссссс | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |

Note: Similar table will be produced for Table 14.3.1.14.

Data source: 16.2.23 Listing of adverse events

Table 14.3.1.15 Duration of the last recurrence of SAEs

| | | Treatment | | | |
|---|---|---|---|---|---|
| | | DFP+DFP DFO+DFP | | | |
| SAE | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value<br>(T-test) |
| Ccccc | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Ccccc | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| •••• | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Ccccc | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |

Note: Similar table will be produced for Table 14.3.1.16.

Data source: 16.2.23 Listing of adverse events

Table 14.3.2.1 Temperature at each assessment

| | D | FP+DFP | P+DFP DFO+DFP | | |
|---|---|---|---|---|---|
| Visit | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value (T-test) |
| Baseline | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 1 | xxx | xx.x ± xx.x<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 2 | XXX | xx.x ± xx.x<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 3 | XXX | xx.x ± xx.x<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 4 | XXX | xx.x ± xx.x<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 5 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 6 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 7 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 8 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 9 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 10 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 11 | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 12 | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 15 | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 18 | XXX | $xx.x \pm xx.x$ $(xx, xx)$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 21 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Month 24 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Month 27 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |

| | Treatment | | | | |
|---|---|---|---|---|---|
| | Б | FP+DFP | ] | DFO+DFP | |
| Month 30 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Month 33 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Month 36 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |

Note: Similar tables will be produced for resting heart rate, respiration, systolic and diastolic blood pressures.

Table 14.3.2.2 Change in temperature from baseline to each follow-up assessment

| | | Tr | eatment | | |
|---|---|---|---|---|---|
| | | DFP+DFP | DFO+DFP | | |
| Visit | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD (Min, Max) | P-value (T-test) |
| Month 1 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 2 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 3 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 4 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 5 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 6 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 7 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 8 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 9 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 10 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 11 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |

| | | Tr | eatment | | |
|---|---|---|---|---|---|
| | I | OFP+DFP | I | DFO+DFP | |
| Month 12 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 15 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Month 18 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Month 21 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Month 24 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 27 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 30 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 33 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 36 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |

Note: Similar tables will be produced for resting heart rate, respiration, systolic and diastolic blood pressures.

Table 14.3.3.1 Weight (kg) at each assessment

| Table 14.5.3 | | | | | |
|---|---|---|---|---|---|
| | Б | FP+DFP | D | FO+DFP | |
| Visit | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value<br>(T-test) |
| Baseline | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 1 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxx |
| Month 2 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 3 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 4 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 5 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 6 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 7 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 8 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 9 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 10 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 11 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 12 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 15 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 18 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 21 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 24 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 27 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |

| - 1 | | L.T | | | |
|---|---|---|---|---|---|
| | D | FP+DFP | D | FO+DFP | |
| Month 30 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | Xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 33 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | Xxx | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Month 36 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | Xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |

Table 14.3.3.2 Change in weight from baseline to last assessment

| | | Treat | | |
|---|---|---|---|---|
| | | DFP+DFP | DFO+DFP | |
| | N | xxx | xxx | P-value<br>(T-test) |
| Change in | Baseline | xxx.x ± xxx.x<br>(xxx, xxx) | xxx.x ± xxx.x<br>(xxx, xxx) | 0.xxxx |
| weight (kg)<br>Mean ± SD | Last assessment | xxx.x ± xxx.x<br>(xxx, xxx) | $xxx.x \pm xxx.x$ $(xxx, xxx)$ | 0.xxxx |
| (Min, Max) | Change at last assessment | xxx.x ± xxx.x<br>(xxx, xxx) | $xxx.x \pm xxx.x$<br>(xxx, xxx) | 0.xxxx |

Table 14.3.3.1 Height (cm) at each assessment

| | Г | FP+DFP | DF | FO+DFP | |
|---|---|---|---|---|---|
| Visit | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD (Min, Max) | P-value<br>(T-test) |
| Baseline | xxx | $xxx \pm xxx$<br>(xxx, xxx) | XXX | xxx ± xxx<br>(xxx, xxx) | 0.xxxx |
| Month 6 | xxx | xxx ± xxx<br>(xxx, xxx) | XXX | xxx ± xxx<br>(xxx, xxx) | 0.xxxx |
| Month 12 | xxx | xxx ± xxx<br>(xxx, xxx) | xxx | xxx ± xxx<br>(xxx, xxx) | 0.xxxx |
| Month 24 | xxx | xxx ± xxx<br>(xxx, xxx) | xxx | xxx ± xxx<br>(xxx, xxx) | 0.xxxx |
| Month 36 | xxx | xxx ± xxx<br>(xxx, xxx) | xxx | xxx ± xxx<br>(xxx, xxx) | 0.xxxx |

Data source: 16.2.5 Listing of vital signs including height and weight

Table 14.3.3.4 Change in height from baseline to last assessment

| | | Treat | | |
|---|---|---|---|---|
| | | DFP+DFP | DFO+DFP | |
| , | N | xxx | xxx | P-value<br>(T-test) |
| Change in | Baseline | xxx.x ± xxx.x<br>(xxx, xxx) | xxx.x ± xxx.x<br>(xxx, xxx) | 0.xxxx |
| height (cm) Mean ± SD (Min, Max) | Last assessment | xxx.x ± xxx.x<br>(xxx, xxx) | xxx.x ± xxx.x<br>(xxx, xxx) | 0.xxxx |
| | Change at last assessment | xxx.x ± xxx.x<br>(xxx, xxx) | xxx.x ± xxx.x<br>(xxx, xxx) | 0.xxxx |

Table 14.3.4.1 Concomitant medications

| = 0 | Trea | Treatment |
|---|---|---|
| | DFP+DFP | DFO+DFP |
| | (N=xxx) | (N=xxx) |
| | Exposure (patient-years): x.xx | Exposure (patient-years): x.xx |
| | Total Patients Reporting: xx | Total Patients Reporting: xx |
| Preferred<br>Name | n Patients (%) | n Patients (%) |
| Ccccc | x (x.x) | x (x.x) |
| Ccccc | x (x.x) | x (x.x) |
| Ccccc | x (x.x) | x (x.x) |

Data source: 16.2.21 Listing of medication

Table 14.3.5.1 Heart rate of 12-lead ECG at each assessment

| | | DFP+DFP | | DFO+DFP | |
|---|---|---|---|---|---|
| Visit | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value<br>(T-test) |
| Baseline | xxx | $xxx \pm xxx$<br>(xxx, xxx) | xxx | xxx ± xxx<br>(xxx, xxx) | 0.xxxx |
| Month 6 | XXX | $xxx \pm xxx$<br>(xxx, xxx) | xxx | $xxx \pm xxx$ $(xxx, xxx)$ | NA |
| Month 12 | XXX | $xxx \pm xxx$ $(xxx, xxx)$ | xxx | $xxx \pm xxx$<br>(xxx, xxx) | 0.xxxx |
| Month 24 | xxx | $xxx \pm xxx$<br>(xxx, xxx) | xxx | xxx ± xxx<br>(xxx, xxx) | 0.xxxx |
| Month 36 | xxx | xxx ± xxx<br>(xxx, xxx) | xxx | xxx ± xxx<br>(xxx, xxx) | NA |

Note: Similar tables will be produced for PR (ms), QRS (ms), QT (ms), QTcF (ms), and QTcB (ms), respectively.

Data source: 16.2.7 Listing of 12-lead electrocardiogram

Table 14.3.5.2 Change in heart rate of 12-lead ECG at each follow-up assessment

| | Γ | )FP+DFP | DI | FO+DFP | |
|---|---|---|---|---|---|
| Visit | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD (Min, Max) | P-value<br>(T-test) |
| Month 6 | xxx | $xxx \pm xxx$ $(xxx, xxx)$ | xxx | xxx ± xxx<br>(xxx, xxx) | NA |
| Month 12 | xxx | $xxx \pm xxx$<br>(xxx, xxx) | xxx | xxx ± xxx<br>(xxx, xxx) | 0.xxxx |
| Month 24 | xxx | xxx ± xxx<br>(xxx, xxx) | xxx | xxx ± xxx<br>(xxx, xxx) | 0.xxxx |
| Month 36 | xxx | $xxx \pm xxx$<br>(xxx, xxx) | xxx | xxx ± xxx<br>(xxx, xxx) | NA |

Note: Similar tables will be produced for PR (ms), QRS (ms), QT (ms), QTcF (ms), and QTcB (ms),

respectively.

Data source: 16.2.7 Listing of 12-lead electrocardiogram

Table 14.3.5.3 Shift table for clinically significant abnormality for 12-lead ECG: DFP+DFP group

| | | La | Last Assessment | |
|---|---|---|---|---|
| | n (%) | Normal | Abnormal | P-value<br>(McNemar's test) |
| Baseline | Normal | xx (xx) | xx (xx) | 0.xxxx |
| | Abnormal | xx (xx) | xx (xx) | |

P-value = Data source: 16.2.7 Listing of 12-lead electrocardiogram

Table 14.3.5.4 Shift table for clinically significant abnormality for 12-lead ECG: DFO+DFP group

| | | La | ast Assessment | |
|----------|----------|---------|----------------|--------------------------|
| | n (%) | Normal | Abnormal | P-value (McNemar's test) |
| Baseline | Normal | xx (xx) | xx (xx) | 0.xxxx |
| | Abnormal | xx (xx) | xx (xx) | |

P-value = Data source: 16.2.7 Listing of 12-lead electrocardiogram

Table 14.3.6.1.1 Hemoglobin at each assessment

| Hemoglobin | D | FP+DFP | DFO+DFP | | P-value<br>(T-test) |
|---|---|---|---|---|---|
| Visit | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | |
| Baseline | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 1 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 2 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 3 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 4 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 5 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 6 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 7 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 8 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 9 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 10 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 11 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 12 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 13 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 14 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 15 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 16 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 17 | XXX | $\begin{array}{c} (xx, xx) \\ xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} (xx, xx) \\ xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |

| | | 4 | | | |
|---|---|---|---|---|---|
| Hemoglobin | DFP+DFP | | oglobin DFP+DFP DFO | | DFO+DFP |
| Week 18 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 19 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 20 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Week 21 | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | XXX | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Week 22 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Week 23 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Week 24 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 25 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 26 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 27 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 28 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 29 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 30 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 31 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 32 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 33 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 34 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 35 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 36 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |

| | | <i>u</i> | | | |
|---|---|---|---|---|---|
| Hemoglobin | D | FP+DFP | DI | DFO+DFP | |
| Week 37 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 38 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 39 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 40 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 41 | xxx | xx.x ± xx.x<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 42 | XXX | xx.x ± xx.x<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 43 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 44 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 45 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 46 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 47 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 48 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 49 | xxx | xx.x ± xx.x<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 50 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 51 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 12 | xxx | xx.x ± xx.x<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 15 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 18 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 21 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |

| - | | | | | |
|---|---|---|---|---|---|
| Hemoglobin | DFP+DFP | | DFO+DFP | | P-value<br>(T-test) |
| Month 24 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 27 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 30 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx,x \pm xx.x \\ (xx,xx) \end{array}$ | 0.xxxx |
| Month 33 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 36 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |

Note: Similar tables will be produced for total white blood cell (WBC), absolute neutrophil count (ANC), and platelets.

Data source: 16.2.9 Listing of hematology

Table 14.3.6.1.2 Change in hemoglobin at each follow-up assessment

| Hemoglobin | DFP+DFP DFO+DFP | | P-value<br>(T-test) | | |
|---|---|---|---|---|---|
| Visit | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | |
| Week 1 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 2 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 3 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 4 | xxx | xx.x ± xx.x<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 5 | xxx | xx.x ± xx.x<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 6 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 7 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 8 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |

| | | Trea | atment | | |
|------------|-----|-----------------|--------|-----------------|----------|
| Hemoglobin | Г | FP+DFP | DI | FO+DFP | P-value |
| | | | | | (T-test) |
| Week 9 | XXX | $xx.x \pm xx.x$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 10 | XXX | $xx.x \pm xx.x$ | xxx | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 11 | XXX | $XX.X \pm XX.X$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 12 | XXX | $XX.X \pm XX.X$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 13 | XXX | $xx.x \pm xx.x$ | xxx | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 14 | XXX | $xx.x \pm xx.x$ | xxx | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 15 | XXX | $xx.x \pm xx.x$ | xxx | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 16 | XXX | XX.X ± XX.X | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 17 | XXX | $xx.x \pm xx.x$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 18 | XXX | XX.X ± XX.X | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 19 | XXX | $xx.x \pm xx.x$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 20 | XXX | $xx.x \pm xx.x$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 21 | XXX | $xx.x \pm xx.x$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 22 | XXX | $xx.x \pm xx.x$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 23 | XXX | $xx.x \pm xx.x$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 24 | XXX | $xx.x \pm xx.x$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 25 | XXX | $xx.x \pm xx.x$ | xxx | $xx.x \pm xx.x$ | 0.xxxx |
| | - | (xx, xx) | | (xx, xx) | |
| Week 26 | XXX | $xx.x \pm xx.x$ | XXX | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | |
| Week 27 | XXX | $xx.x \pm xx.x$ | xxx | $xx.x \pm xx.x$ | 0.xxxx |
| | | (xx, xx) | | (xx, xx) | _ |

| | □ 7·4 <sub>1</sub> | _ | | | |
|---|---|---|---|---|---|
| Hemoglobin | D: | DFP+DFP DFO+DFP P-<br>(T | | DFO+DFP | |
| Week 28 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 29 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 30 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 31 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 32 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 33 | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 34 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 35 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 36 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 37 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 38 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 39 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 40 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 41 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 42 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 43 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 44 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 45 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 46 | xxx | $\begin{array}{c} (XX, XX) \\ XX.X \pm XX.X \\ (XX, XX) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |

| | = 2 | | | | |
|---|---|---|---|---|---|
| Hemoglobin | Γ | )FP+DFP | Di | FO+DFP | P-value<br>(T-test) |
| Week 47 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 48 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 49 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Week 50 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Week 51 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 12 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 15 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 18 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 21 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 24 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 27 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 30 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 33 | XXX | $xx.x \pm xx.x$ $(xx, xx)$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 36 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |

Note: Similar tables will be produced for total white blood cell (WBC), absolute neutrophil count (ANC), and platelets.

Data source: 16.2.9 Listing of hematology

Table 14.3.6.1.3 Shift table for hemoglobin in abnormal range at baseline vs last assessment:

DFP+DFP group

| | n (%) | Low | Normal | High | P-value<br>(McNemar's test) |
|---|---|---|---|---|---|
| | Low | xx (xx) | xx (xx) | xx (xx) | |
| Baseline | Normal | xx (xx) | xx (xx) | xx (xx) | 0.xxxx |
| | High | xx (xx) | xx (xx) | xx (xx) | |

Note: Similar tables will be produced for total white blood cell (WBC), absolute neutrophil count

(ANC), and platelets.

Data source: 16.2.9 Listing of hematology

Table 14.3.6.1.4 Shift table for hemoglobin in abnormal range at baseline vs last assessment: DFO+DFP group

| = = | n (%) | Low | Normal | High | P-value<br>(McNemar's test) |
|---|---|---|---|---|---|
| | Low | xx (xx) | xx (xx) | xx (xx) | |
| Baseline | Normal | xx (xx) | xx (xx) | xx (xx) | 0.xxxx |
| | High | xx (xx) | xx (xx) | xx (xx) | |

Note: Similar tables will be produced for total white blood cell (WBC), absolute neutrophil count

(ANC), and platelets.

Data source: 16.2.9 Listing of hematology

Table 14.3.6.2.1 Total protein at each assessment

| | Γ | FP+DFP | D | DFO+DFP | |
|---|---|---|---|---|---|
| Visit | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value<br>(T-test) |
| Baseline | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 1 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 2 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 3 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Month 4 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 5 | xxx | | | 0.xxxx | |
| Month 6 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Month 7 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Month 8 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Month 9 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 10 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 11 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 12 | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 18 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $\begin{array}{c} (xx, xx) \\ xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 24 | XXX | $xx.x \pm xx.x$ $(xx, xx)$ | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 30 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $XX.X \pm XX.X$ $(XX, XX)$ | 0.xxxx |
| Month 36 | XXX | $xx.x \pm xx.x$ $(xx, xx)$ | XXX | (xx, xx)<br>(xx, xx) | 0.xxxx |

Note: Similar tables will be produced for GGT, lactate dehydrogenase (LDH), sodium, potassium, chloride, glucose (fasting at screening visit only), total, direct and indirect bilirubin, AST, ALT, albumin; blood urea nitrogen, calcium, creatinine, uric acid, alkaline phosphatase, and amylase. Data source: 16.2.12 Listing of chemistry

Table 14.3.6.2.2 Change in total protein at each follow-up assessment

| | D | FP+DFP | DI | FO+DFP | |
|---|---|---|---|---|---|
| Visit | N Mean ± SD (Min, Max) | | N | Mean ± SD<br>(Min, Max) | P-value<br>(T-test) |
| Month 1 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 2 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 3 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | xxx | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Month 4 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 5 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Month 6 | XXX | $xx.x \pm xx.x$ $(xx, xx)$ | XXX | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Month 7 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 8 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 9 | XXX | $xx.x \pm xx.x$<br>(xx, xx) | XXX | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |
| Month 10 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Month 11 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | XXX | xx.x ± xx.x<br>(xx, xx) | 0.xxxx |
| Month 12 | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $xx.x \pm xx.x$<br>(xx, xx) | 0.xxxx |
| Month 18 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\(xx, xx) \end{array}$ | 0.xxxx |
| Month 24 | xxx | xx.x ± xx.x<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 30 | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |
| Month 36 | xxx | $xx.x \pm xx.x$<br>(xx, xx) | xxx | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | 0.xxxx |

Note: Similar tables will be produced for GGT, lactate dehydrogenase (LDH), sodium, potassium, chloride, glucose (fasting at screening visit only), total, direct and indirect bilirubin, AST, ALT, albumin; blood urea nitrogen, calcium, creatinine, uric acid, alkaline phosphatase, and amylase. Data source: 16.2.12 Listing of chemistry

Table 14.3.6.2.3 Shift table for total protein in abnormal range at baseline vs last assessment: DFP+DFP group

| | n (%) | Low | Normal | High | P-value<br>(McNemar's test) |
|---|---|---|---|---|---|
| | Low | xx (xx) | xx (xx) | xx (xx) | |
| Baseline | Normal | xx (xx) | xx (xx) | xx (xx) | 0.xxxx |
| | High | xx (xx) | xx (xx) | xx (xx) | |

Note: Similar tables will be produced for GGT, lactate dehydrogenase (LDH), sodium, potassium, chloride, glucose (fasting at screening visit only), total, direct and indirect bilirubin, AST, ALT, albumin; blood urea nitrogen, calcium, creatinine, uric acid, alkaline phosphatase, and amylase. Data source: 16.2.12 Listing of chemistry

Table 14.3.6.2.4 Shift table for total protein in abnormal range at baseline vs last assessment: DFO+DFP group

| | n (%) | Low | Normal | High | P-value<br>(McNemar's test) |
|---|---|---|---|---|---|
| | Low | xx (xx) | xx (xx) | xx (xx) | |
| Baseline | Normal | xx (xx) | xx (xx) | xx (xx) | 0.xxxx |
| | High | xx (xx) | xx (xx) | xx (xx) | |

Note: Similar tables will be produced for GGT, lactate dehydrogenase (LDH), sodium, potassium, chloride, glucose (fasting at screening visit only), total, direct and indirect bilirubin, AST, ALT, albumin; blood urea nitrogen, calcium, creatinine, uric acid, alkaline phosphatase, and amylase. Data source: 16.2.12 Listing of chemistry

Table 14.3.6.3.1 HIV Antibody at each assessment

| | DF | P+DFP | DFC | )+DFP | P-value<br>(Fisher's<br>exact test) |
|---|---|---|---|---|---|
| | N | Positive<br>n (%) | N | Positive n (%) | |
| Baseline | xxx | xx (xx) | xxx | xx (xx) | 0xxxx |
| Month 6 | xxx | xx (xx) | xxx | xx (xx) | 0.xxxx |
| Year 1 | xxx | xx (xx) | xxx | xx (xx) | 0.xxxx |
| Year 3 | xxx | xx (xx) | xxx | xx (xx) | 0.xxxx |

Note: Similar tables will be produced for Hepatitis B and C.

Data source: 16.2.13 Listing of serology

Table 14.3.7.1 Female patients with positive pregnancy test during the study

| | Treatment | |
|---|---|---|
| Pregnancy test: Positive | DFP+DFP | DFO+DFP |
| Patient ID | xxxxxx<br>xxxxxx<br>xxxxxx | xxxxxx<br>xxxxxx<br>xxxxxx<br>xxxxxx |
| | ••••• | ***** |

Data source: 16.2.14 Listing of pregnancy

Table 14.4.1 The number and percent of patients who had compliance  $\leq$ 80% or  $\geq$ 120% during the study

| | Г | FP+DFP | D | FO+DFP | |
|---|---|---|---|---|---|
| Compliance | N | Percent | N | Percent | P-value<br>(Fisher's exact<br>test) |
| < 80% | xx | xx.x% | xx | xx.x% | 0.xxxx |
| > 120% | xx | xx.x% | xx | xx.x% | 0.xxxx |

Data source: 16.2.19 Listing of compliance

Table 14.5.1 Overall mean of transfusional iron input (mg/kg/day) during the study

| | 1 (8-8-1), 1-1-18 | | | | |
|---|---|---|---|---|---|
| | | Treat | | | |
| | Γ | DFP+DFP | DFO+DFP | | P-value<br>(T-test) |
| | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD (Min, Max) | |
| Overall mean of transfusional iron input (mg/kg/day) | xxx | xx.x ± xx.x<br>(xx, xx) | xxx | $xx.x \pm xx.x$ $(xx, xx)$ | 0.xxxx |

Data source: 16.2.26 Listing of transfusion information

Table 14.6.1 Overall mean of total daily dose

| | | Treatment | | |
|---|---|---|---|---|
| | DFP+DFP DFO+DFI | | | |
| | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) |
| Overall mean of total daily dose (mg/kg/day) | XXX | $\begin{array}{c} xx.x \pm xx.x \\ (xx, xx) \end{array}$ | xxx | xx.x ± xx.x<br>(xx, xx) |

Data source: 16.2.24 Listing of exposure